CLINICAL TRIAL: NCT04714424
Title: Comparing Vision Tests Integrated Into a Virtual Reality Technology Against Its Currently Used Analogues
Brief Title: Comparing Vision Tests in a Virtual Reality Headset to Existing Analogues
Acronym: RTS1
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, James Chelnis, Assistant Clinical Professor, MD, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 19-03280
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Ptosis; Macular Degeneration; Ametropia
Keywords: Vision screening; Virtual reality; Field test; Visual acuity; Contrast sensitivity
MeSH Terms: conditions — Blepharoptosis; Macular Degeneration; Refractive Errors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Participants undergoing vision exams
  Interventions: Device: Virtual Reality Headset

INTERVENTIONS:
Device: Virtual Reality Headset — Virtual reality (VR) - a 3-D reality right in a headset
  Other Names: Vive Pro

SUMMARY:
The purpose of this study is to compare the results of vision tests that are algorithmically derived and delivered through a virtual reality headset with those delivered through the existing technology standards (eg. Humphrey for field tests). Tests that the researchers will be conducting include vision field perimetry, Amsler, acuity chart, contrast- sensitivity and currently used office tests.

DETAILED DESCRIPTION:
Virtual reality (VR) constructs a 3-D reality right in a headset and the researchers are studying with what degree of accuracy it can be use to recreate vision tests that are used by eye doctors to screen and diagnose patients. VR provides advantages that could be used to improve eye care once the technology is tested and compared to the currently used vision tests - such as limiting the costs, duration and tedium associated with existing forms of vision screening tests. By doing so, the researchers hope to expand access to eye care by lowering the cost burden associated with vision tests. In this study, the research team will have subjects go through the VR versions of the test that are used in practice, and analyze their results in comparison to one another. After informed consent is obtained, the research team will collect subject demographic information (date of birth, gender, ethnicity, race) and clinically relevant medical history. Afterward, the research team will proceed to the virtual reality tests: vision field perimetry, Amsler, Snellen chart, contrast- sensitivity and currently used office tests. The participants will undergo all the tests, VR and non-VR, which will be delivered in a randomized order. The entire sequence will last 30 minutes to one hour for a single test. The VR component will last about 5 minutes, this being the only addition to the scheduled vision tests. The sequence of VR / non VR testing will be randomized. Based on the previous studies that compared Humphrey MATRIX visual field and Swedish Interactive algorithm, the effect size is determined to be at least 30 subjects, and the goal is to reach N=1,000 participants.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of any race who are at least 18 years of age and can understand and provide verbal and written informed consent are eligible for this study.

Exclusion Criteria:

* Patients who have had intraocular surgery less than six months ago,
* Potential contraindication for visual field test that include anxiety disorder, pregnancy, seizure disorder,cardiac pacemaker or another implantable device, severe vertigo or balance issues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from New York Eye and Ear Infirmary.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Vision Field Perimetry | Day 1
  Vision field perimetry will me measured using Humphrey Vision Field Analyzer and a VR equivalent software.
Acuity | Day 1
  Acuity will be measured using Tumbling E and LogMAR tests and a VR version of those tests.
Contrast | Day 1
  Contrast sensitivity will be measured using the Pelli-Robson test and a VR version of the test.
Color vision | Day 1
  Color vision will be measured by Ishihara plates and a VR version of the test.

SECONDARY OUTCOMES:
Patient Satisfaction Survey | Day 1
  The survey consists of Likert scale questions to understand the patient's experience with the VR and analogues. The scale is evaluated from 1 to 5, with 1 meaning "very poor" and 5 meaning "very good". Score for each section (HVFA and VR) is 3 to 15. Total scale is 6 to 30, with higher score indicating more satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: James Chelnis, MD, Principal Investigator — New York Eye and Ear Infirmary of Mount Sinai
Locations (1):
- New York Eye & Ear Infirmary of Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. Data available on specific request and will be shared securely as CSV.

REFERENCES:
- [Background] Heijl A, Patella VM, Chong LX, Iwase A, Leung CK, Tuulonen A, Lee GC, Callan T, Bengtsson B. A New SITA Perimetric Threshold Testing Algorithm: Construction and a Multicenter Clinical Study. Am J Ophthalmol. 2019 Feb;198:154-165. doi: 10.1016/j.ajo.2018.10.010. Epub 2018 Oct 16. PMID 30336129
- [Background] Kimura T, Matsumoto C, Nomoto H. Comparison of head-mounted perimeter (imo(R)) and Humphrey Field Analyzer. Clin Ophthalmol. 2019 Mar 14;13:501-513. doi: 10.2147/OPTH.S190995. eCollection 2019. PMID 30936681
- [Background] Lowry EA, Hou J, Hennein L, Chang RT, Lin S, Keenan J, Wang SK, Ianchulev S, Pasquale LR, Han Y. Comparison of Peristat Online Perimetry with the Humphrey Perimetry in a Clinic-Based Setting. Transl Vis Sci Technol. 2016 Jul 19;5(4):4. doi: 10.1167/tvst.5.4.4. eCollection 2016 Jul. PMID 27486554
- [Background] Phu J, Khuu SK, Yapp M, Assaad N, Hennessy MP, Kalloniatis M. The value of visual field testing in the era of advanced imaging: clinical and psychophysical perspectives. Clin Exp Optom. 2017 Jul;100(4):313-332. doi: 10.1111/cxo.12551. Epub 2017 Jun 22. PMID 28640951
- [Background] Prema R, George R, Hemamalini A, Sathyamangalam Ve R, Baskaran M, Vijaya L. Comparison of Humphrey MATRIX and Swedish interactive threshold algorithm standard strategy in detecting early glaucomatous visual field loss. Indian J Ophthalmol. 2009 May-Jun;57(3):207-11. doi: 10.4103/0301-4738.49395. PMID 19384015
- [Background] Scarfe P, Glennerster A. Using high-fidelity virtual reality to study perception in freely moving observers. J Vis. 2015;15(9):3. doi: 10.1167/15.9.3. PMID 26161632
- [Background] Sharma AK, Goldberg I, Graham SL, Mohsin M. Comparison of the Humphrey swedish interactive thresholding algorithm (SITA) and full threshold strategies. J Glaucoma. 2000 Feb;9(1):20-7. doi: 10.1097/00061198-200002000-00005. PMID 10708227
- [Background] Barbour KE, Helmick CG, Boring M, Brady TJ. Vital Signs: Prevalence of Doctor-Diagnosed Arthritis and Arthritis-Attributable Activity Limitation - United States, 2013-2015. MMWR Morb Mortal Wkly Rep. 2017 Mar 10;66(9):246-253. doi: 10.15585/mmwr.mm6609e1. PMID 28278145
- [Background] Beard C. Muller's superior tarsal muscle: anatomy, physiology, and clinical significance. Ann Plast Surg. 1985 Apr;14(4):324-33. doi: 10.1097/00000637-198504000-00005. PMID 3994278
- [Background] Collin JR, Beard C, Wood I. Experimental and clinical data on the insertion of the levator palpebrae superioris muscle. Am J Ophthalmol. 1978 Jun;85(6):792-801. doi: 10.1016/s0002-9394(14)78107-3. PMID 98045
- [Background] Cosh S, Carriere I, Daien V, Tzourio C, Delcourt C, Helmer C. Sensory loss and suicide ideation in older adults: findings from the Three-City cohort study. Int Psychogeriatr. 2019 Jan;31(1):139-145. doi: 10.1017/S104161021800056X. Epub 2018 May 25. PMID 29798742
- [Background] DeBuc DC. The Role of Retinal Imaging and Portable Screening Devices in Tele-ophthalmology Applications for Diabetic Retinopathy Management. Curr Diab Rep. 2016 Dec;16(12):132. doi: 10.1007/s11892-016-0827-2. PMID 27841014
- [Background] Lee CS, Morris A, Van Gelder RN, Lee AY. Evaluating Access to Eye Care in the Contiguous United States by Calculated Driving Time in the United States Medicare Population. Ophthalmology. 2016 Dec;123(12):2456-2461. doi: 10.1016/j.ophtha.2016.08.015. Epub 2016 Sep 12. PMID 27633646
- [Background] Goh RLZ, Kong YXG, McAlinden C, Liu J, Crowston JG, Skalicky SE. Objective Assessment of Activity Limitation in Glaucoma with Smartphone Virtual Reality Goggles: A Pilot Study. Transl Vis Sci Technol. 2018 Jan 23;7(1):10. doi: 10.1167/tvst.7.1.10. eCollection 2018 Jan. PMID 29372112
- [Background] Hootman JM, Helmick CG, Barbour KE, Theis KA, Boring MA. Updated Projected Prevalence of Self-Reported Doctor-Diagnosed Arthritis and Arthritis-Attributable Activity Limitation Among US Adults, 2015-2040. Arthritis Rheumatol. 2016 Jul;68(7):1582-7. doi: 10.1002/art.39692. PMID 27015600
- [Derived] Cheng CP, Serafini RA, Labkovich M, Warburton AJ, Navarro V, Shaik N, Reddy H, Chelnis JG. Clinical report: Virtual reality enables comparable contrast sensitivity measurements to in-office testing (pilot study). Optom Vis Sci. 2024 Feb 1;101(2):124-128. doi: 10.1097/OPX.0000000000002107. Epub 2024 Jan 16. PMID 38408310